CLINICAL TRIAL: NCT03053115
Title: Combined Replacement Therapy With Levothyroxine and Liothyronine in Thyroidectomized Patients: Effects on Peripheral Tissues. A Prospective, Randomized, Controlled, Double-blind Study
Brief Title: Combined Replacement Therapy With Levothyroxine and Liothyronine in Thyroidectomized Patients
Acronym: LEVOLIO
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Azienda USL Modena (Other)
Responsible Party: Principal Investigator, Manuela Simoni, Director of the Unit of Endocrinology, Azienda USL Modena
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EudraCT: 2016-000687-41
Record Dates: First submitted 2016-11-25; First posted 2017-02-14 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Hypothyroidism
Keywords: thyroid; levothyroxine; combined therapy
MeSH Terms: conditions — Hypothyroidism; Thyroid Diseases | interventions — Triiodothyronine; Thyroxine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CASES (Experimental): treatment with levothyroxine and liothyronine
  Interventions: Drug: Liothyronine; Drug: Levothyroxin
- CONTROLS (Active Comparator): treatment with levothyroxine and placebo
  Interventions: Drug: Levothyroxin; Drug: Placebos

INTERVENTIONS:
Drug: Liothyronine — Cases will take liothyronine drops in the morning and two hours after dinner
  Arms: CASES
Drug: Levothyroxin — Both cases and controls will take levothyroxine in the morning (entire dose for controls, reduced dose for cases)
Drug: Placebos — Controls will take placebo two hours after dinner
  Arms: CONTROLS

SUMMARY:
The aim of the study is to evaluate the peripheral tissue response to the combined administration of levothyroxine (LT4) and liothyronine (LT3) in hypothyroid patients with residual thyroid function virtually absent (thyroidectomized). Cases will be treated with LT4+LT3, at personalized doses according to clinical guidelines and respecting the circadian rhythmicity of LT3 and the physiological T3/T4 ratio. Controls will be treated with LT4 and placebo. Treatment duration: 24 weeks.

The primary endpoint will be the peripheral effect of thyroid hormones. The secondary endpoints are bone and metabolic modifications, and changes in quality of life. Moreover any changes of outcomes related to polymorphisms of genes involved in thyroid hormones metabolism will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years
* capable of consent
* able to fill in a questionnaire in italian
* thyroidectomized
* serum thyroglobulin levels below 0.2 ng/ml and antibodies anti-thyroglobulin undetectable (below normal range)
* well treated taking stable doses of levothyroxine in tablets, in the previous 3 months

Exclusion Criteria:

* TSH suppressive therapy
* pregnancy
* cardiac arrhythmias
* severe liver, kidney or bone diseases
* ongoing steroids treatment
* ongoing or in the previous 12 months treatment with bone anti-resorptive, amiodarone, colestyramine or iron.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2021-09-05 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
change from baseline SHBG serum levels at 12 and 24 weeks (nmol/L) | baseline and then repeated at 12 weeks and 24 weeks
  change from baseline SHBG serum levels at 12 and 24 weeks (nmol/L)

SECONDARY OUTCOMES:
BMI (kg/m2) | baseline and then repeated at 6, 12 weeks and 24 weeks
  body mass index
quality of life changes | baseline and then repeated at 12 weeks and 24 weeks
  score at validated questionnaires
change from baseline TSH serum levels at 12 and 24 weeks (microIU/ml) | baseline and then repeated at 12 weeks and 24 weeks
  change from baseline TSH serum levels at 12 and 24 weeks (microIU/ml)
change from baseline free triiodothyronine (fT3) serum levels at 12 and 24 weeks (pmol/L) | baseline and then repeated at 12 weeks and 24 weeks
  change from baseline free triiodothyronine (fT3) serum levels at 12 and 24 weeks (pmol/L)
change from baseline free levothyroxine (fT4) serum levels at 12 and 24 weeks (pmol/L) | baseline and then repeated at 12 weeks and 24 weeks
  change from baseline free levothyroxine (fT4) serum levels at 12 and 24 weeks (pmol/L)
change from baseline total cholesterol serum levels at 12 and 24 weeks (mg/dl) | baseline and then repeated at 12 weeks and 24 weeks
  change from baseline total cholesterol serum levels at 12 and 24 weeks (mg/dl)
change from baseline HDL cholesterol serum levels at 12 and 24 weeks (mg/dl) | baseline and then repeated at 12 weeks and 24 weeks
  change from baseline HDL cholesterol serum levels at 12 and 24 weeks (mg/dl)
change from baseline triglycerides serum levels at 12 and 24 weeks (mg/dl) | baseline and then repeated at 12 weeks and 24 weeks
  change from baseline triglycerides serum levels at 12 and 24 weeks (mg/dl)
change from baseline C-terminal telopeptide of type 1 collagen at 12 and 24 weeks (ng/dl) | baseline and then repeated at 12 weeks and 24 weeks
  change from baseline C-terminal telopeptide of type 1 collagen at 12 and 24 weeks (ng/dl)
change from baseline Osteocalcin at 12 and 24 weeks (ng/mL) | baseline and then repeated at 12 weeks and 24 weeks
  change from baseline Osteocalcin at 12 and 24 weeks (ng/mL)
change from baseline Bone alkaline phosphatase at 12 and 24 weeks (µg/L) | baseline and then repeated at 12 weeks and 24 weeks
  change from baseline Bone alkaline phosphatase at 12 and 24 weeks (µg/L)

CONTACTS AND LOCATIONS:
Locations (1):
- AziendaUSLModena, Modena, Italy